CLINICAL TRIAL: NCT05849350
Title: Effects of Pilates Training and Protein Supplementation on Body Composition, Performance, and Biochemical Indices
Brief Title: Protein Supplementation in Pilates Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PilatesProtein1
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Exercise Training; Dietary Supplements
MeSH Terms: interventions — Whey Proteins; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein (Experimental): Participants will receive a whey protein supplement.
  Interventions: Dietary Supplement: Whey protein
- Maltodextrin (Placebo Comparator): Participants will receive an isocaloric maltodextrin supplement.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Whey protein — Intake of whey protein
  Arms: Protein
Dietary Supplement: Maltodextrin — Intake of maltodextrin
  Arms: Maltodextrin

SUMMARY:
Pilates training, a type of mind and body exercise that focuses on muscle strength and flexibility, has become increasingly popular in recent years. Research has shown that Pilates could be an effective exercise form to improve body composition, particularly in obese individuals, while beneficial effects on flexibility, muscular strength, and muscular endurance have also been observed in young and older adults. It is well documented that protein supplementation can augment the effects of resistance training on body composition and performance. While there is an abundance of studies investigating the effect of protein supplements on adaptations to resistance exercise, there is a knowledge gap regarding their effectiveness in Pilates training.

The aim of this research is to investigate the effects of protein supplementation, compared to placebo (maltodextrin) on body composition, performance, and biochemical indices in healthy young and middle-aged, eumenorrheic (regular menstrual cycle) women who perform Pilates. Participants will be randomly assigned to receive either 0.6 g of whey protein or maltodextrin per kg body weight per day for 10 weeks. Participants will be asked to avoid modifying their dietary habits for the duration of the study to limit the effect of diet on the measured parameters. To check for this, participants will record their diet for 3 days (2 weekdays and one weekend day) on the first, middle, and last weeks of the intervention. Dietary records will then be analyzed. Pilates classes will be performed at least two times per week, while specialized Pilates equipment (Reformer or Cadillac) will be used according to the Pilates principles. The duration of each workout will be set at around 50 min.

Participants will undergo measurements of body composition, core muscle endurance, and joint flexibility at the beginning and end of the study. In addition, hematologic parameters, clinical chemistry parameters, hormones, and plasma amino acids will be measured. All these outcome measures will be compared between the whey protein and maltodextrin groups to determine the effectiveness of protein supplementation in Pilates training.

ELIGIBILITY:
Inclusion Criteria:

* Eumenorrheic (regular menstrual cycle) women
* Regular Pilates training (at least 2 times a week, 50 min each session, for the past 4 months), as assessed by gym records or questionnaires
* Mixed isoenergetic diet for the past 4 months

Exclusion Criteria:

* Any musculoskeletal injuries that could interfere with training
* Chronic disease
* Milk allergy
* Pregnancy, lactation, or planning a pregnancy within the duration of the study
* Regular use of prescription medicine or supplements that might affect muscle function or recovery over the past month
* Intermittent or religious fasting
* Any vegetarian, ketogenic or protein diet

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Lean mass and fat mass pre-supplementation | Within one week before the beginning of supplementation.
  Lean mass and fat mass of the whole body and its parts (arms, legs, trunk) will be assessed by dual X-ray absorptiometry. Whole body lean, dry lean and fat mass will also be assessed by multifrequency bioelectrical impedance analysis.
Lean mass and fat mass post-supplementation | Within one week after the end of supplementation.
  Lean mass and fat mass of the whole body and its parts (arms, legs, trunk) will be assessed by dual X-ray absorptiometry. Whole body lean, dry lean and fat mass will also be assessed by multifrequency bioelectrical impedance analysis.
Bone mineral density pre-supplementation | Within one week before the beginning of supplementation.
  Bone mineral density of the whole body and its parts (arms, legs, trunk) will be assessed by dual X-ray absorptiometry.
Bone mineral density post-supplementation | Within one week after the end of supplementation.
  Bone mineral density of the whole body and its parts (arms, legs, trunk) will be assessed by dual X-ray absorptiometry.
Bone mineral content pre-supplementation | Within one week before the beginning of supplementation.
  Bone mineral content of the whole body and its parts (arms, legs, trunk) will be assessed by dual X-ray absorptiometry.
Bone mineral content post-supplementation | Within one week after the end of supplementation.
  Bone mineral content of the whole body and its parts (arms, legs, trunk) will be assessed by dual X-ray absorptiometry.
Bone area pre-supplementation | Within one week before the beginning of supplementation.
  Bone area of the whole body and its parts (arms, legs, trunk) will be assessed by dual X-ray absorptiometry.
Bone area post-supplementation | Within one week after the end of supplementation.
  Bone area of the whole body and its parts (arms, legs, trunk) will be assessed by dual X-ray absorptiometry.
Body fat % and lean % pre-supplementation | Within one week before the beginning of supplementation.
  Body fat as a % of total body weight will be assessed by dual X-ray absorptiometry and multifrequency bioelectrical impedance analysis. Lean as a % of total body weight will be assessed by multifrequency bioelectrical impedance analysis.
Body fat % and lean % post-supplementation | Within one week after the end of supplementation.
  Body fat as a % of total body weight will be assessed by dual X-ray absorptiometry and multifrequency bioelectrical impedance analysis. Lean as a % of total body weight will be assessed by multifrequency bioelectrical impedance analysis.
Body weight pre-supplementation | Within one week before the beginning of supplementation.
  Body weight will be measured with an electronic scale to the nearest 0.1 kg
Body weight post-supplementation | Within one week after the end of supplementation.
  Body weight will be measured with an electronic scale to the nearest 0.1 kg
Waist and hip circumferences pre-supplementation | Within one week before the beginning of supplementation.
  Waist and hip circumferences will be measured with a non-extendable tape
Waist and hip circumferences post-supplementation | Within one week after the end of supplementation.
  Waist and hip circumferences will be measured with a non-extendable tape
Joint flexibility pre-supplementation | Within one week before the beginning of supplementation.
  Joint flexibility will be assessed through the sit and reach test.
Joint flexibility post-supplementation | Within one week after the end of supplementation.
  Joint flexibility will be assessed through the sit and reach test.
Core muscle endurance pre-supplementation | Within one week before the beginning of supplementation.
  Core muscle endurance (trunk flexor, trunk lateral right, trunk lateral left, and trunk extensors) will be assessed through the McGill's torso muscular endurance test battery.
Core muscle endurance post-supplementation | Within one week after the end of supplementation.
  Core muscle endurance (trunk flexor, trunk lateral right, trunk lateral left, and trunk extensors) will be assessed through the McGill's torso muscular endurance test battery.
Plasma glucose, total cholesterol, HDL cholesterol, LDL cholesterol, and triacylglycerols pre-supplementation | Within one week before the beginning of supplementation.
  Plasma glucose, total cholesterol, HDL cholesterol, LDL cholesterol, and triacylglycerols (all in mg/dL) will be measured by chemiluminescence in an automated analyzer.
Plasma glucose, total cholesterol, HDL cholesterol, LDL cholesterol, and triacylglycerols post-supplementation | Within one week after the end of supplementation.
  Plasma glucose, total cholesterol, HDL cholesterol, LDL cholesterol, and triacylglycerols (all in mg/dL) will be measured by chemiluminescence in an automated analyzer.
Plasma amino acid profile pre-supplementation | Within one week before the beginning of supplementation.
  Plasma amino acid profile (that is, the concentration of each individual amino acid) will be determined by liquid chromatography-mass spectrometry.
Plasma amino acid profile post-supplementation | Within one week after the end of supplementation.
  Plasma amino acid profile (that is, the concentration of each individual amino acid) will be determined by liquid chromatography-mass spectrometry.

SECONDARY OUTCOMES:
Full blood count pre-supplementation | Within one week before the beginning of supplementation.
  Full blood count will be performed by flow cytometry
Full blood count post-supplementation | Within one week after the end of supplementation.
  Full blood count will be performed by flow cytometry
Plasma enzymes pre-supplementation | Within one week before the beginning of supplementation.
  Creatine kinase and γ-glutamyltransferase (both in U/L) will be measured by chemiluminescence in an automated analyzer
Plasma enzymes post-supplementation | Within one week after the end of supplementation.
  Creatine kinase and γ-glutamyltransferase (both in U/L) will be measured by chemiluminescence in an automated analyzer
Cortisol pre-supplementation | Within one week before the beginning of supplementation.
  Plasma Cortisol (μg/dL) will be measured by immunoluminescence in an automated analyzer.
Cortisol post-supplementation | Within one week after the end of supplementation.
  Plasma Cortisol (μg/dL) will be measured by immunoluminescence in an automated analyzer.
Progesterone and testosterone pre-supplementation | Within one week before the beginning of supplementation.
  Plasma progesterone and testosterone (both in ng/dL) will be measured by immunoluminescence in an automated analyzer.
Progesterone and testosterone post-supplementation | Within one week after the end of supplementation.
  Plasma progesterone and testosterone (both in ng/dL) will be measured by immunoluminescence in an automated analyzer.
Estradiol pre-supplementation | Within one week before the beginning of supplementation.
  Plasma estradiol (pg/mL) will be measured by immunoluminescence in an automated analyzer.
Estradiol post-supplementation | Within one week after the end of supplementation.
  Plasma estradiol (pg/mL) will be measured by immunoluminescence in an automated analyzer.
Plasma urea and creatinine pre-supplementation | Within one week before the beginning of supplementation.
  Plasma urea and creatinine (both in mg/dL) will be measured by chemiluminescence in an automated analyzer.
Plasma urea and creatinine post-supplementation | Within one week after the end of supplementation.
  Plasma urea and creatinine (both in mg/dL) will be measured by chemiluminescence in an automated analyzer.
Total body water %, intracellular water %, and extracellular water % pre-supplementation | Within one week before the beginning of supplementation.
  Total body water, intracellular water, and extracellular water (all as % of total body weight) will be assessed by multifrequency bioelectrical impedance analysis.
Total body water %, intracellular water %, and extracellular water % post-supplementation | Within one week after the end of supplementation.
  Total body water, intracellular water, and extracellular water (all as % of total body weight) will be assessed by multifrequency bioelectrical impedance analysis.
Total body water, intracellular water, and extracellular water pre-supplementation | Within one week before the beginning of supplementation.
  Total body water, intracellular water, and extracellular water (all in Lt) will be assessed by multifrequency bioelectrical impedance analysis.
Total body water, intracellular water, and extracellular water post-supplementation | Within one week after the end of supplementation.
  Total body water, intracellular water, and extracellular water (all in Lt) will be assessed by multifrequency bioelectrical impedance analysis.
Body mass index (BMI) pre-supplementation | Within one week before the beginning of supplementation
  BMI will be calculated by divinding weight by height squared.
Body mass index (BMI) post-supplementation | Within one week after the end of supplementation.
  BMI will be calculated by divinding weight by height squared.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Evaluation of Human Biological Performance, Thessaloniki, Greece